CLINICAL TRIAL: NCT00601627
Title: Phase II Study of Panitumumab, Chemotherapy, and External Beam Radiation in Patients With Locally Advanced Pancreatic Cancer
Brief Title: Panitumumab, Chemotherapy, and External-Beam Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N064A; NCI-2009-01088 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000584104 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2008-01-18; First posted 2008-01-28 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Panitumumab; Capecitabine; Fluorouracil; Gemcitabine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Panitumumab (Experimental): Chemotherapy concurrent with radiation: Radiation 5 days per week for 5½ weeks; Panitumumab on days 1, 15, and 29 of radiation therapy 5-fluorouracil (5FU) continuous infusion, starting on day 1 and through last day of radiation.
  4-6 weeks after completion of radiation therapy: Gemcitabine on days 1, 8, and 15 of each cycle, for 3 cycles; Panitumumab on days 1 and 15 of each cycle, for 3 cycles. Maintenance therapy: Panitumumab on days 1 and 15 of each cycle, for 6 cycles.
  Interventions: Biological: panitumumab; Drug: capecitabine; Drug: fluorouracil; Drug: gemcitabine hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: panitumumab
Drug: capecitabine
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Monoclonal antibodies, such as panitumumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as fluorouracil, capecitabine, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. External-beam radiation therapy uses high-energy x-rays to kill tumor cells. Panitumumab may also stop the growth of pancreatic cancer by blocking blood flow to the tumor and make tumor cells more sensitive to radiation therapy. Giving panitumumab together with chemotherapy and radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving panitumumab together with chemotherapy and external-beam radiation therapy works in treating patients with locally advanced pancreatic cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To evaluate the 1-year survival rate in patients with locally advanced pancreatic cancer treated with panitumumab and continuous infusion fluorouracil administered concurrently with external-beam radiotherapy followed by gemcitabine and panitumumab.

Secondary

* To determine overall survival, time to disease progression, confirmed response rate, duration of response, and time to treatment failure in patients treated with this regimen.
* To determine adverse events in patients treated with this regimen.

OUTLINE:

* Panitumumab and chemoradiotherapy : Patients undergo external-beam radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33, and 36-38. Patients also receive panitumumab IV over 1 hour on days 1, 15, and 29 and fluorouracil IV continuously over 24 hours daily OR oral capecitabine twice daily beginning on day 1 and continuing through the last day of radiotherapy.
* Panitumumab and chemotherapy: Beginning 4-6 weeks after completion of panitumumab and chemoradiotherapy, patients receive panitumumab IV over 1 hour on days 1 and 15 and gemcitabine IV over 30 minutes on days 1, 8, and 15. Treatment repeats every 28 days for 3 courses. Patients then proceed to maintenance therapy.
* Maintenance therapy: Patients receive panitumumab IV over 1 hour on days 1 and 15. Treatment repeats every 28 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed every 3 months for 2 years and then every 6 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed unresectable adenocarcinoma of the pancreas

  * Including subtotal resection and gross residual disease

    * No microscopic residual disease only
* Measurable disease is not required
* Disease is encompassable within standard radiotherapy fields for pancreatic cancer
* No evidence of metastatic disease outside of the planned radiotherapy field
* No cystadenocarcinoma of the pancreas or pancreatic tumors of neuroendocrine origin
* No distant metastases (i.e., liver or lung metastases or peritoneal spread)
* No history or known presence of CNS metastases

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* ANC ≥ 1,500/mm³
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/mm³
* Total bilirubin ≤ 3 times upper limit of normal (ULN)* NOTE: *Biliary stent placement or surgical bypass should be considered prior to treatment if impending bile duct obstruction by tumor
* AST ≤ 3 times ULN
* Creatinine ≤ 2.0 times ULN
* Magnesium normal
* Willing to return to an North Central Cancer Treatment Group (NCCTG) institution for follow-up
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 6 months after treatment with panitumumab
* No prior or concurrent malignancy unless disease-free ≥ 3 years except for non-melanoma skin cancer, carcinoma in situ of the cervix, or organ confined prostate cancer with Gleason score < 7
* No nausea or vomiting > grade 1
* No uncontrolled intercurrent illness including, but not limited to, any the following:

  * Ongoing or active infection
  * Psychiatric illness or social situations that would limit compliance with study requirements
* No New York Heart Association clinically significant cardiovascular disease ≥ grade 2, including any of the following within the past year:

  * Myocardial infarction
  * Unstable angina
  * Symptomatic congestive heart failure
  * Serious, uncontrolled cardiac arrhythmia
* No known HIV positivity
* No known hepatitis C virus or acute or chronic active hepatitis B infection
* Adequate oral nutrition

PRIOR CONCURRENT THERAPY:

* More than 21 days since prior laparotomy
* No prior anti-epidermal growth factor receptor (EGFR) antibody therapy (e.g., cetuximab)
* No prior small molecule EGFR inhibitors (e.g., gefitinib, erlotinib, or lapatinib)
* No prior radiotherapy that would overlap with planned radiotherapy fields
* No prior or other concurrent chemotherapy
* No prior or other concurrent biologic therapy
* More than 4 weeks since prior and no concurrent or planned participation in another experimental drug study except studies with specific interventions intended to treat rashes associated with EGFR agents (e.g., N05C4)
* No concurrent enteral hyperalimentation
* No concurrent chronic immunosuppressive agents (e.g., methotrexate, cyclosporine, or corticosteroids)
* No concurrent colony-stimulating factors during the first course of therapy
* No other concurrent immunotherapy or radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-06; Primary Completion 2011-07 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George Kim, MD, Study Chair — Mayo Clinic
Locations (281):
- United States (281):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Saint Francis/Mount Sinai Regional Cancer Center at Saint Francis Hospital and Medical Center, Hartford, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Illinois CancerCare - Bloomington, Bloomington, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Illinois CancerCare - Canton, Canton, Illinois
  - Illinois CancerCare - Carthage, Carthage, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Illinois CancerCare - Eureka, Eureka, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare - Galesburg, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Illinois CancerCare - Havana, Havana, Illinois
  - Mason District Hospital, Havana, Illinois
  - Illinois CancerCare - Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare - Macomb, Macomb, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Moline, Illinois
  - Illinois CancerCare - Monmouth, Monmouth, Illinois
  - OSF Holy Family Medical Center, Monmouth, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Illinois CancerCare - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Illinois CancerCare - Pekin, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare - Peru, Peru, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Illinois CancerCare - Princeton, Princeton, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Illinois CancerCare - Spring Valley, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart Clinic, LLC, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology-Oncology, PC - South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - South Bend Clinic, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Bettendorf, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, Clive, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - McCreery Cancer Center at Ottumwa Regional, Ottumwa, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Liberal, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Dickinson County Healthcare System, Iron Mountain, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital - Monroe, Monroe, Michigan
  - Mercy General Health Partners, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Lakeside Cancer Specialists, PLLC, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Duluth Clinic Cancer Center - Duluth, Duluth, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller - Dwan Medical Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Wood County Oncology Center, Bowling Green, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - North Coast Cancer Care - Clyde, Clyde, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Toledo Clinic - Oregon, Oregon, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Geisinger Hazleton Cancer Center, Hazleton, Pennsylvania
  - Geisinger Medical Group - Scenery Park, State College, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - Fredericksburg Oncology, Incorporated, Fredericksburg, Virginia
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Marshfield Clinic - Chippewa Center, Chippewa Falls, Wisconsin
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Holy Family Memorial Medical Center Cancer Care Center, Manitowoc, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Marshfield Clinic at Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

REFERENCES:
- [Derived] Halfdanarson TR, Foster NR, Kim GP, Haddock MG, Dakhil SR, Behrens RJ, Alberts SR. N064A (Alliance): Phase II Study of Panitumumab, Chemotherapy, and External Beam Radiation in Patients with Locally Advanced Pancreatic Adenocarcinoma. Oncologist. 2022 Jul 5;27(7):534-e546. doi: 10.1093/oncolo/oyac002. PMID 35285484

RESULTS

PARTICIPANT FLOW:
Groups:
- Panitumumab: Chemotherapy concurrent with radiation:
  Radiation 5 days per week for 5½ weeks; 6 mg/kg Panitumumab on days 1, 15, and 29 of radiation therapy 225 mg/m^2 per day 5-fluorouracil (5FU) continuous infusion, starting on day 1 and through last day of radiation.
  4-6 weeks after completion of radiation therapy: 1000 mg/m^2 Gemcitabine on days 1, 8, and 15 of each cycle, for 3 cycles; 6 mg/kg Panitumumab on days 1 and 15 of each cycle, for 3 cycles.
  Maintenance therapy:
  6 mg/kg Panitumumab on days 1 and 15 of each cycle, for 6 cycles.
Period: Overall Study
Arm/Group | Panitumumab
Started | 51
Completed | 51
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All patients were included in this analysis.
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
Age, Continuous [Median (Full Range); unit: years] | 65 [43 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 51

OUTCOME MEASURES:

1. Primary Outcome: One Year Survival Rate
Description: The proportion of successes will be estimated by the number of successes divided by the total number of evaluable patients. Confidence intervals for the true success proportion will be calculated according to the exact binomial method.
Time Frame: Baseline to 12 months
Population: All patients were evaluable for this endpoint.
Measure: Number (95% Confidence Interval); unit: proportion of patients
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
proportion of patients | 0.502 [0.354 to 0.632]

2. Secondary Outcome: Overall Survival
Description: Survival time is defined as the time from registration to death due to any cause. The distribution of survival time will be estimated using the method of Kaplan-Meier
Time Frame: baseline to 2 years
Population: All patients were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
months | 12.1 [6.8 to 15.1]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival is defined as the time from registration to the earliest documented evidence of disease progression.
Time Frame: baseline to 2 years
Population: All patients were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
months | 7.4 [3.7 to 8.6]

4. Secondary Outcome: Confirmed Response Rate
Description: A confirmed tumor response is defined to be a complete response (CR) or partial response (PR) noted as the objective status on 2 consecutive evaluations at least 4 weeks apart according to the Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1.
  A complete response is defined as the disappearance of all target and non-target lesions.
  A partial response is defined as at least a 30% decrease in the sum of the longest diameter (LD) of the target lesion from baseline.
  Confirmed tumor response will be evaluated using the first 6 cycles of treatment.
Time Frame: baseline to 2 years
Population: All patients were analyzed for this endpoint.
Measure: Number (95% Confidence Interval); unit: rate of confirmed response
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
rate of confirmed response | 0.059 [0.012 to 0.162]

5. Secondary Outcome: Duration of Response
Description: Duration of response is defined for all evaluable patients who have achieved an objective response as the date at which the patient's earliest best objective status is first noted to be either a CR or PR to the earliest date progression is documented.
Time Frame: baseline to 2 years
Population: Too few patients reported a confirmed response to provide meaningful information into the duration of response.
Arm/Group | Panitumumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Time to Treatment Failure
Description: Time to treatment failure is defined to be the time from the date of registration to the date at which the patient is removed from treatment due to progression, adverse events, or refusal. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: baseline to 2 years
Population: All patients were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panitumumab
Number analyzed (Participants) | 51
months | 2.71 [1.54 to 4.24]

ADVERSE EVENTS:
Groups:
- Panitumumab: 6 mg/kg Panitumumab on days 1 and 15 of each cycle, for 6 cycles.
Arm/Group | Panitumumab
Serious Adverse Events (participants affected / at risk) | 29/51
Other Adverse Events (participants affected / at risk) | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab (N=51)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 7 (8)
Duodenal obstruction (Gastrointestinal disorders) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 3 (4)
Esophageal stenosis (Gastrointestinal disorders) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 9 (10)
Small intestine ulcer (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (8)
Fever (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disease (Hepatobiliary disorders) | 1 (1)
Biliary tract infection (Infections and infestations) | 2 (2)
Bladder infection (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 3 (5)
Creatinine increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 4 (5)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (5)
Anorexia (Metabolism and nutrition disorders) | 4 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 11 (11)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Panitumumab (N=51)
Hemoglobin decreased (Blood and lymphatic system disorders) | 41 (126)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 11 (16)
Ascites (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 30 (64)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 21 (33)
Flatulence (Gastrointestinal disorders) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 16 (23)
Nausea (Gastrointestinal disorders) | 40 (83)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 31 (52)
Chest pain (General disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Edema limbs (General disorders) | 4 (4)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 47 (137)
Fever (General disorders) | 7 (7)
Abdominal infection (Infections and infestations) | 3 (8)
Catheter related infection (Infections and infestations) | 1 (1)
Esophageal infection (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infectious colitis (Infections and infestations) | 1 (1)
Opportunistic infection (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (7)
Alkaline phosphatase increased (Investigations) | 5 (8)
Aspartate aminotransferase increased (Investigations) | 8 (10)
Bilirubin increased (Investigations) | 5 (6)
Creatinine increased (Investigations) | 5 (7)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 32 (79)
Lymphocyte count decreased (Investigations) | 10 (17)
Neutrophil count decreased (Investigations) | 19 (36)
Platelet count decreased (Investigations) | 28 (63)
Weight loss (Investigations) | 9 (13)
Anorexia (Metabolism and nutrition disorders) | 43 (86)
Blood bicarbonate decreased (Metabolism and nutrition disorders) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 7 (9)
Dehydration (Metabolism and nutrition disorders) | 9 (13)
Serum albumin decreased (Metabolism and nutrition disorders) | 6 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 7 (9)
Serum magnesium decreased (Metabolism and nutrition disorders) | 29 (87)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 4 (4)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (4)
Taste alteration (Nervous system disorders) | 4 (8)
Depression (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (27)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 (29)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (8)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 (8)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 3 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 8 (19)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (57)
Rash acneiform (Skin and subcutaneous tissue disorders) | 35 (84)
Rash desquamating (Skin and subcutaneous tissue disorders) | 21 (43)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (5)
Hot flashes (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 3 (5)
Thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less